CLINICAL TRIAL: NCT03114319
Title: An Open-label, Multi-center, Phase I, Dose Finding Study of Oral TNO155 in Adult Patients With Advanced Solid Tumors
Brief Title: Dose Finding Study of TNO155 in Adult Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons and not due to any safety concerns
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTNO155X2101; 2023-508925-29-00 (Other: EU CTIS)
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Advanced EGFR Mutant Non Small Cell LungCancer (NSCLC); KRAS G12-mutant NSCLC; Esophageal Squamous Cell Cancer (SCC); Head/Neck SCC; Melanoma; Advanced Gastrointestinal Stromal Tumors (GIST); Advanced NRAS/BRAFT wt Cutaneous Melanoma
Keywords: TNO155; SHP2; advanced solid tumor; NSCLC; HNSCC; Esophageal SCC; Melanoma; EGFR; KRAS G12C; GIST; PTPN11; cancers with a mass; bulky tumor; nodule; lump; advanced solid malignancies
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Melanoma; Squamous Cell Carcinoma of Head and Neck; Noonan Syndrome | interventions — nazartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNO155 (Experimental): TNO155 for oral administration
  Interventions: Drug: TNO155
- TNO155 in combination with EGF816 (nazartinib) (Experimental): TNO155 in combination with EGF816 (nazartinib) in patients with advanced EGFR mutant NSCLC
  Interventions: Drug: TNO155 in combination with EGF816 (nazartinib)

INTERVENTIONS:
Drug: TNO155 — TNO155 for oral administration
  Arms: TNO155
Drug: TNO155 in combination with EGF816 (nazartinib) — TNO155 for oral administration; EGF816 (nazartinib) for oral administration
  Arms: TNO155 in combination with EGF816 (nazartinib)

SUMMARY:
The purpose of this first in human (FIH) trial was to characterize the safety and tolerability of the SHP2 inhibitor TNO155 alone and in combination with EGF816 (nazartinib) and identify a recommended dose for future studies in adult patients with advanced solid tumors in selected indications.

DETAILED DESCRIPTION:
This study has been designed as a Phase I, open-label, dose finding study with a dose escalation part and a dose expansion part in adult patients with selected advanced solid tumors. The study treatment, TNO155 alone or in combination with EGF816 (nazartinib), was taken until the patient experienced unacceptable toxicity, progressive disease and/or treatment was discontinued at the discretion of the investigator or the patient or due to withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign the ICF and able to comply with the study visit schedule and the other protocol requirements.
2. Patient (male or female) ≥18 years of age willing to agree to not father a child/become pregnant and comply with effective contraception criteria.
3. Must have progressed following standard therapy, or for whom, in the opinion of the Investigator, no effective standard therapy exists, is tolerated or is appropriate.
4. ECOG (Eastern cooperative oncology group) performance status ≤2

   Additional criteria only appying to TNO155 in combination with EGF816 (nazartinib):
5. Patients must be screened for Hepatitis B virus and Hepatitis C virus

Exclusion Criteria:

1. Tumors harboring known activating KRAS, NRAS, HRAS, BRAF or PTPN11 (SHP2) mutations. (Exceptions are KRAS G12-mutant NSCLC's)
2. History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO.
3. Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
4. Clinically significant cardiac disease.
5. Active diarrhea or inflammatory bowel disease
6. Insufficient bone marrow function
7. Insufficient hepatic and renal function.

   Additional criteria only appying to TNO155 in combination with EGF816 (nazartinib):
8. Patients with a known history of human immunodeficiency virus (HIV) seropositivity.
9. Patients receiving concomitant immunosuppressive agents or chronic corticosteroids use at the time of study entry.
10. Patients who have undergone a bone marrow or solid organ transplant
11. Patients with a history or presence of interstitial lung disease or interstitial pneumonitis
12. Bullous and exfoliative skin disorders at screening of any grade
13. Presence of clinically significant ophthalmological abnormalities that might increase the risk of corneal epithelial injury

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events | up to 5 years; at least once per treatment cycle
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms and cardiac biomarkers
Number of participants with dose limiting toxicities | up to 28-day cycle
  Incidence and nature of dose limiting toxicities (DLTs) in the dose escalation part. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle (either 21 days or 28 days, depending on the cohort's treatment schedule) with TNO155 or with TNO155 in combination with EGF816 (nazartinib)
Number of participants with dose interruptions and reductions | Up to 5 years
  Assessment of tolerability. For patients who do not tolerate the protocol-specified dosing schedule, dose adjustments may be permitted in order to allow patients to continue the study treatment
Dose intensity of study drugs | Up to 5 years
  Dose intensity is computed as the ratio of actual cumulative dose received to actual duration of exposure

SECONDARY OUTCOMES:
Overall response rate (ORR) per RECIST v1.1 | From start of treatment for 60 months
  ORR is the proportion of patients with a best overall response of Complete Response (CR) or Partial response (PR)
Disease control rate (DCR) per RECIST v1.1 | From start of treatment for 60 months
  DCR is the proportion of patients with a best overall response of CR or PR or stable disease (SD)
Progression-free survival (PFS) per RECIST v1.1 | Up to 5 years
  PFS is the time from date start of treatment to the date of event defined as the first documented progression or death due to any cause
Duration of response (DOR) per RECIST v1.1 | Up to 5 years
  DOR is the time from first documented response (PR or CR) to the date of first documented disease progression or death due to any cause
Change from baseline in DUSP6 in tumor samples | At screening and between Cycle 1 and Cycle 3. One cycle=either 21 days or 28 days, depending on the cohort's treatment schedule.
  Dual Specificity Phosphatase 6 (DUSP6) mRNA levels assessed in paired tumor biopsy samples by quantitative polymerase chain reaction (qPCR)
Area under the plasma concentration-time curve (AUC) of study drugs | From pre-dose up to 48 hours post-dose on Cycle 1 Day 1 and from pre-dose up to 24 hours post-dose on Cycle 1 Day 14. One cycle=21 days or 28 days, depending on the dosing schedule.
  Pharmacokinetic (PK) parameters calculated based on the plasma concentrations versus time profiles by using non-compartmental methods
Peak plasma concentration (Cmax) of study drugs | From pre-dose up to 48 hours post-dose on Cycle 1 Day 1 and from pre-dose up to 24 hours post-dose on Cycle 1 Day 14. One cycle=21 days or 28 days, depending on the dosing schedule.
  PK parameters calculated based on the plasma concentrations versus time profiles by using non-compartmental methods
Time to reach peak plasma concentration (Tmax) of study drugs | From pre-dose up to 48 hours post-dose on Cycle 1 Day 1 and from pre-dose up to 24 hours post-dose on Cycle 1 Day 14. One cycle=21 days or 28 days, depending on the dosing schedule.
  PK parameters calculated based on the plasma concentrations versus time profiles by using non-compartmental methods
Apparent terminal elimination half-life of study drugs | From pre-dose up to 48 hours post-dose on Cycle 1 Day 1 and from pre-dose up to 24 hours post-dose on Cycle 1 Day 14. One cycle=21 days or 28 days, depending on the dosing schedule.
  PK parameters calculated based on the plasma concentrations versus time profiles by using non-compartmental methods

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (4):
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Memorial Sloane Ketterin Cancer Ctr, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Kobe, Japan
- Netherlands (2):
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, Amsterdam
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (3):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No